CLINICAL TRIAL: NCT04506190
Title: A Prospective Multicenter Study to Evaluate the Perioperative Outcomes of Robotic-assisted Revisional Bariatric Surgery
Brief Title: Prospective Robotic-assisted Revisional Bariatric Study
Status: Completed | Type: Observational
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: ISI-dVBR-002
Record Dates: First submitted 2020-08-05; First posted 2020-08-10 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Bariatric Surgery Candidate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Robotic-assisted revisional bariatric surgery: Subjects who undergo robotic-assisted revisional bariatric surgery
  Interventions: Procedure: Revisional bariatric surgery

INTERVENTIONS:
Procedure: Revisional bariatric surgery — Subjects who undergo revisional bariatric surgery

SUMMARY:
Very few studies have compared robotic-assisted (RRBS) versus laparoscopic revisional bariatric surgeries (LRBS). To date, there has not been a prospective study comparing the perioperative outcomes of patients undergoing robotic-assisted and laparoscopic revisional bariatric surgery. This study aims to enroll patients undergoing RRBS and LRBS and evaluate the outcomes through 45 days, including the perioperative period. We hypothesize that RRBS may be associated with lower rates of perioperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years or older at the time of consent
2. Subject has a history of prior bariatric surgery
3. Subject's revisional procedure will be either laparoscopic revisional bariatric surgery (LRBS) or robotic-assisted revisional bariatric surgery (RRBS)
4. Subject undergoes revisional bariatric surgery that is applicable to study

Exclusion Criteria:

1. Subject is undergoing a primary bariatric procedure
2. Subject has undergone more than one previous bariatric procedure
3. Subject's revisional bariatric procedure is an emergent procedure
4. Subject is contraindicated for general anesthesia or surgery
5. Subject is unable to comply with the follow-up visit schedule
6. Subject is pregnant or suspects pregnancy
7. Subject is mentally handicapped or has a psychological disorder or severe systemic illness that would preclude compliance with study requirements or ability to provide informed consent
8. Subject belonging to other vulnerable population, e.g, prisoner or ward of the state

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have had one previous bariatric surgery, are undergoing a revisional bariatric surgery applicable to this study, and who are deemed qualified by study inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Rate of conversions | During the surgical procedure
  Conversions is defined as RRBS to LRBS or open revisional bariatric surgery, and LRBS to open revisional bariatric surgery

SECONDARY OUTCOMES:
Postoperative rate of anastomotic leak | 45 days after date of procedure
  Anastomotic leak is defined as a leak of luminal contents from a surgical join

CONTACTS AND LOCATIONS:
Locations (1):
- Orlando Health, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
All individual participant data that underlie results in a publication